CLINICAL TRIAL: NCT00899808
Title: Molecular and Genetic Markers in the Local-regional Management of Patients Undergoing Radiation Therapy
Brief Title: Molecular Markers and Genetic Markers in Patients Undergoing Radiation Therapy for Cancer
Status: Withdrawn | Type: Observational
Why Stopped: not "applicable clinical trial"
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 000609; P30CA072720 (NIH); CDR0000592887; CINJ-IRB-0220060141
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Hematopoietic/Lymphoid Cancer; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; hematopoietic/lymphoid cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at molecular markers and genetic markers in patients undergoing radiation therapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine local-regional control in patients undergoing radiation therapy for cancer, as a function of expression of specific molecular/genetic markers.

Secondary

* Determine complications of radiation therapy for patients undergoing radiation therapy for cancer.

OUTLINE: Previously collected tissue samples are analyzed using immunohistochemical staining and other molecular/genetic study methods to detect markers, including p53, cyclin D1, HER-2-neu, bcl-2/BAX, and EGFR. Patient charts are also reviewed with emphasis on local-regional relapse.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Undergoing radiation therapy for malignant disease

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing radiation therapy for malignant disease will be eligible for these studies. Initially we will focus on specific disease sites, such as breast, prostate and lung, but ultimately we will expand this to include any disease site. Patients who met standard criteria for radiation therapy but ultimately did not receive radiation therapy will be used as a control arm if needed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Haffty, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey- Robert Wood Johnson Medical School
Locations (1):
- Rutgers Cancer Institute of New Jersey - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States